CLINICAL TRIAL: NCT02681224
Title: TR-987 vs. Placebo Following Fractionated CO2 Laser Resurfacing of the Chest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TR987-2013-01
Record Dates: First submitted 2016-02-08; First posted 2016-02-12 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Exposure Laser

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Active Product with Occlusion (Active Comparator): TR987 Gel with Silon Bandage
  Interventions: Other: TR987 Gel with Silon Bandage
- Active Product without Occlusion (Active Comparator): TR987 without Silon Bandage
  Interventions: Other: TR987 without Silon Bandage
- Placebo Gel with Occlusion (Placebo Comparator): Placebo Gel with Silon Bandage
  Interventions: Other: Placebo Gel with Silon Bandage
- Placebo Gel without Occlusion (Placebo Comparator): Placebo Gel without Silon Bandage
  Interventions: Other: Placebo Gel without Silon Bandage

INTERVENTIONS:
Other: TR987 Gel with Silon Bandage — Novel healing gel with occlusive dressing
  Arms: Active Product with Occlusion
Other: TR987 without Silon Bandage — Novel healing gel without occlusive dressing
  Arms: Active Product without Occlusion
Other: Placebo Gel with Silon Bandage — Placebo gel with occlusive dressing
  Arms: Placebo Gel with Occlusion
Other: Placebo Gel without Silon Bandage — Placebo Gel without occlusive dressing
  Arms: Placebo Gel without Occlusion

SUMMARY:
A single site, double-blind, randomized, placebo-controlled, clinical study comparing the difference between a novel healing gel and a placebo gel on post laser-resurfacing chests.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, chest clinical study with a single study site. Forty subjects will receive fractionated CO2 laser resurfacing of the chest. . Immediately following the procedure (Day 0), postoperative gel randomized to the chest (TR-987 or placebo), will be applied with a thickness of 1-2 mm by a non-blinded coordinator, along with a split-chest Silon TSR bandage. Subjects will return for follow up on Day 1, with the gel and split chest Silon TSR© bandages applied by non-blinded coordinator during visit, with further follow-up on Days 6, 8, 10, 13 and 28. Both subjects and evaluating investigator will be blinded to randomization schedule (performed by an unblinded coordinator). Subject will apply gels and split chest Silon TSR© bandages at home on Days 2, 3 and 4 when not visiting clinic.

ELIGIBILITY:
Inclusion Criteria:

* Females or males in good general health greater than 18 years of age.
* Must be willing to give and sign a HIPPA form, informed consent form, and a photographic release form
* Subject is planning to undergo fractionated CO2 laser resurfacing to the chest
* A potential subject's must exhibit:

  --Skin phototype of Fitzpatrick Type I-IV
* For FEMALE SUBJECT OF CHILDBEARING POTENTIAL, must have had a regular menstrual cycle prior to study entry (a female is considered of childbearing potential unless she is postmenopausal, without a uterus and/or both ovaries, or has had a bilateral tubal ligation) and is willing to use an acceptable form of birth control during the entire course of the study [i.e., acceptable methods of birth control are oral contraceptives, contraceptive patches/rings/implants Norplant®, Depo-Provera®, double-barrier methods (e.g. condoms and spermicide), abstinence and vasectomies of partner with a documented second acceptable method of birth control should the subject become sexually active]. All systemic birth control measures must be in consistent use at least 30 days prior to study participation. Postmenopausal is defined as having the last menstrual cycle in at least 12 months
* Negative urine pregnancy test results at the time of study entry (if applicable)
* Must be willing to comply with study dosing and complete the entire course of the study.

Exclusion Criteria:

* A subject with any UNCONTROLLED systemic disease at the discretion of the Investigator. A potential subject in whom therapy for a systemic disease is not yet stabilized will not be considered for entry into the study
* A subject with a significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study.
* A subject with recently excessive exposure to sunlight or artificial UV light (e.g.: use of tanning beds/booths and/or sunbathing) or expectations of tanning during the time of the study or has used self-tanner within 7 days of study entry.
* A subject with history of or the presence of any skin condition/disease that might interfere with the diagnosis or evaluation of study parameters (i.e., atopic dermatitis, eczema, psoriasis, seborrheic dermatitis) at the discretion of the investigator.
* A subject with an active bacterial, fungal, or viral infection in the treatment area.
* A subject with known allergies or sensitivities to benzocaine, lidocaine, tetracaine, PABA (para-aminobenzoic acid), or other local anesthetics of the amide or ester family sedation medication.
* A subject with known allergy or sensitivity to propylene glycol or any other ingredient of topical TR-987 or placebo.
* A subject receiving any topical products containing alpha-hydroxy acids, salicylic acid, and vitamins C or E (includes derivatives thereof) on the chest within 14 days prior to or during the study period, other than the study products
* A subject receiving any investigational drug and/or has had a microdermabrasion (light or medium skin peel) treatment on their chest within 30 days prior to or during the study period
* A subject using any topical tretinoin product or derivative on their chest within 12 weeks prior to or during the study period
* A subject receiving a chemical peel, any systemic steroids, a non-ablative laser, light or radio frequency treatment and/or has had a Dermabrasion (deep skin peel) or ablative laser treatments on their chest must have discontinued the drug/treatment and/or have completed the treatment or the procedure at least 3 months prior to entering the study.
* A subject with a history of keloids or hypertrophic scars
* A subject that has previously been treated with a systemic retinoid within the past year (e.g., Accutane®, Roche Dermatologics)
* A female subject who is pregnant, nursing an infant or planning a pregnancy during the study [throughout the course of the study, women of child-bearing potential must use reliable forms of contraception (i.e., oral contraceptive, contraceptive patches/rings/implants Norplant®, Depo-Provera®, double-barrier methods (e.g. condoms and spermicide), abstinence, or vasectomies of partner with a documented second acceptable method of birth control should the subject become sexually active].
* Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Rate of Healing | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Mitchel P Goldman, MD, Principal Investigator — Cosmetic Laser Dermatology
Locations (1):
- Cosmetic Laser Dermatology, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No